CLINICAL TRIAL: NCT05066113
Title: Feasibility Study on Radiofrequency-Based Selective Electrothermolysis to Investigate Its Effects on Human Skin
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00112812
Record Dates: First submitted 2021-09-01; First posted 2021-10-04 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Hidradenitis Suppurativa; Healthy Volunteers
Keywords: Radiofrequency-Based Selective Electrothermolysis; Hidradenitis Suppurativa; Healthy volunteers
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Intervention Model Description: Participants will be enrolled to test for the tolerability, safety, and histometric changes in skin-RF interactions in axillary skin. RF-based selective electrothermolysis will be administered to skin of healthy volunteers and Hidradenitis Suppurativa (HS) patients at varying depth, intensity, and time.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Healthy Participants (Experimental): Electrothermolysis treatment using varying levels of RF energies
  Interventions: Device: Radiofrequency-Based treatment

INTERVENTIONS:
Device: Radiofrequency-Based treatment — RF-based treatments use electrothermolysis to deliver heat energy to targeted structures in the skin, such as hair follicles or glands by the use of insulated needles. The investigators will use radio frequency based treatment on a pre-selected skin area (about 3cm x 3cm or 1 ¼ x 1 ¼ inches in size) on either your left or right underarm that is eligible for assessment, study treatment, and biopsy.
  Participants will receive clinical assessments, photography, questionnaires, up to 3 treatments of RF-based selective electrothermolysis to pre-selected areas of the axillary skin, up to 2 4-mm skin biopsies for up to 5 study visits.

SUMMARY:
This research is being done to assess the effect of radiofrequency (RF)-based treatment on skin and skin conditions.

DETAILED DESCRIPTION:
Radiofrequency (RF)-based selective electrothermolysis is an increasingly utilized minimally invasive technology for several dermatologic conditions, such as epilation, acne vulgaris, and skin rejuvenation, with minimal side effects. This procedure targets and destroys selective cutaneous and subcutaneous structures; therefore, allowing greater control and specificity of treatment area and minimizing destruction to surrounding tissue. Here, the investigators propose to utilize this technology on human axillary skin to establish safety and biologic effects of selective electrothermolysis in this particular area of the skin.

The investigators will assess the tolerability, safety, and histometric changes in skin-radiofrequency interactions in the axillary skin of participants. The investigators will collect skin samples from prospective volunteers and assess for biologic effects in human axillary skin after selective electrothermolysis treatment.

During the four months of study period, Participants in the study will receive clinical assessments, photography, questionnaires, up to 3 treatments of RF-based selective electrothermolysis to pre-selected areas of the axillary skin, up to 2 4-mm skin biopsies for up to 5 study visits.

ELIGIBILITY:
Inclusion Criteria:

1. For primary objective: healthy volunteers and HS patients between 22 and 70 years of age.
2. Participants must be healthy enough to undergo multiple skin biopsy in the opinion of the investigator.
3. Participants must provide informed consent.
4. Participants must have the ability and willingness to follow all study procedures, attend scheduled visits, and successfully complete the study.
5. Participants must have the ability to understand and communicate with the investigator.
6. For HS patients, participants will have localized disease to the axillae, mild to moderate severity and no evidence of active infection as assessed by the investigator

Exclusion Criteria:

1. Participants unable to provide informed consent.
2. Recently treated for current skin diseases that would affect clinical evaluation.
3. Known contraindications to selective electrothermolysis treatment.
4. Immunocompromised patients
5. Participants on systemic steroids
6. Participants on immune modulators
7. Participants on blood thinners
8. Participants with bleeding disorders
9. Participants with any active infections or currently treated infections
10. Participants with significant medical history or concurrent illness that the investigator feels is not safe for biopsy or study participation.
11. Noncompliant participants.
12. Pregnant or nursing participants (qualitative human chorionic gonadotropin (hCG) testing will be performed prior to each treatment).
13. Participants with allergy to anesthetics.
14. Participants with a history of keloids or hypertrophic scars within the past 10 years.
15. Participants who have taken oral/topical antihistamines, oral/topical analgesics, and/or other medications that the investigators believe will impact the study.
16. Participants who are currently taking or who have taken in the past 12 months any medications that may impair wound healing, such as systemic retinoids.
17. Participants who cannot undergo motor strength and sensory testing required to assess for adverse events in this study.

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-08-15 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Tolerability of skin-RF interactions in axillary skin | 4 months
  Tolerability will be assessed by number of patients experiencing adverse events grade 2 or higher as defined by the Common Terminology Criteria for Adverse Events.
Safety of skin-RF interactions in axillary skin | 4 months
  Safety will be assessed by number of patients experiencing adverse events grade 2 or higher as defined by the Common Terminology Criteria for Adverse Events.

CONTACTS AND LOCATIONS:
Overall Officials: Noori Kim, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No